CLINICAL TRIAL: NCT06259864
Title: Examining the Efficacy of Mollii Suit in Children With Non-Ambule Cerebral Palsy: A Single Blind Randomized Controlled Study.
Brief Title: Effects of Mollii Suit in Children With Non-Ambule Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kübra Uğurlu, research assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CerebralPalyMolliiSuit
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Mollii Suit; Cerebral Palsy
Keywords: cerebral palsy; mollii suit; spasticity; salivation; constipation; gross motor function; quality of life
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Sialorrhea; Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental treatment program group (Active Comparator): NDT aims to bring the child to the maximum level of independence possible within the limits of age and ability. Treatment sessions are planned for a certain functional result, and the patient's active participation as much as possible is requested. As the child fulfills postural and motor requirements, the physical therapist provides less assistance and less guidance. Positionings supported by auxiliary materials, appropriate hand contacts, correct ways to hold the child, tonus regulation, family education, environmental regulations and goal-oriented quality movement approaches; These are some of the methods used by the NDT approach, which is based on facilitation, stimulation and communication. Neurodevelopmental treatment physiotherapy session for 2 days in a week, over 8 week.
  Interventions: Other: EXOPULSE Mollii Suit method
- Mollii Suit method group (Experimental): The Exopulse Mollii Suit is designed to restore normality and healthy balance of muscle groups in the body. The suite uses one of several different forms of neuromodulation, based on gently stimulating the affected muscle groups with electrical signals. This approach has been shown to help resynchronize muscle signals that have been disrupted due to spasticity and muscle groups that may have stopped working together. 58 electrodes embedded in the suit send mild and imperceptible impulses to both tense and spastic muscles and the weakened muscles that balance them. These stimulations not only relax tense muscles and reactivate weak ones, but also restore the natural balance of the group and help the body move as it should. Children will wear the outfit twice a week for 8 weeks and each session will last 60 minutes. During this practice, children will also receive NDT twice a week.
  Interventions: Other: EXOPULSE Mollii Suit method

INTERVENTIONS:
Other: EXOPULSE Mollii Suit method — EXOPULSE Mollii Suit method, one of the newest rehabilitation technology products, is a non-invasive neuromodulation approach with a garment that covers the whole body and electrodes placed inside. Designed to improve motor function by reducing spasticity and pain, the method is based on the principle of reciprocal inhibition, which occurs by stimulating the antagonist of a spastic muscle at low frequencies and intensities.

SUMMARY:
The aim of our study is to examine the effectiveness of the Mollii Suit application on gross motor function, spasticity, postural control, upper extremity skills, selective motor control, daily living activities, quality of life, pain, sleep, constipation and drooling problems in non-ambulatory individuals with cerebral palsy (CP).

DETAILED DESCRIPTION:
Our study includes children diagnosed with spastic type cerebral palsy at GMFCS level 4 or 5 who applied to the Developmental Physiotherapy and Pediatric Rehabilitation Unit of Gazi University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.

After the patients are separated according to the specified exclusion and inclusion criteria, they will be divided into two groups by simple randomization method.

Evaluations will be made before and after treatment. In addition to normal neurodevelopmental therapy (NGT) and Mollii Suit method will be applied 2 days a week. The total duration of treatment will take 8 weeks. Groups; The first group will consist of children with CP who will receive neurodevelopmental treatment.

The second group will consist of children who will receive the Molli Suit method in addition to neurodevelopmental treatment.

ELIGIBILITY:
Inclusion Criteria:

* GMFCS 4 or 5 with spastic cerebral palsy children
* Volunteering to participate in the study

Exclusion Criteria:

* Botulinum toxinA injection in the last 3 months
* Surgical intervention involving the musculoskeletal system in the last 6 months
* Having an invasive medical pump (baclofen, insulin, etc.)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 15 minutes
  GMFM evaluates children's motor activities in 5 different positions called 'lying down and rolling over', 'crawling and kneeling down', 'sitting', 'standing' and 'walking, running, jumping' on a scale of 0-3 (0: unable to initiate movement. 3: independent movement). It is a measurement method that scores.
Modified Tradiue Scale | 5-10 minutes
  Modified Tardiue Scale (MTS) will be used in the evaluation of spasticity. MTS is a method that evaluates the velocity-sensitive nature of spasticity through passive movement. Muscle tone of the ankle plantar flexors will be assessed in both knee flexion and extension. Hamstring spasticity will be tested in the supine position with the pelvic-femoral angle at 90°. After slow and fast stretching of the joint, two values of the angle will be measured according to angle R2 and R1 respectively. R1 is defined as the point in the PEHA at which a catch or clonus is first felt during rapid stretching of the joint, while R2 is defined as the total PEHA of the ankle. R2-R1 represents the dynamic component of spasticity. Spasticity will be measured according to the muscle reaction when stretching as fast as possible and will be graded from 0 to 5.
Modified Ashworth Scale | 5 minutes
  Modified Ashworth Scale (MAS) will be used to evaluate muscle tone. Hamstring and plantar flexor muscle tone evaluation will begin in the supine position, with the head in the midline and the extremities in the resting position, and MAS scores will be determined between 0-4 according to the resistance level of the antagonist muscles during passive movement.
Functional Reach Test | 3 minutes
  Functional Reach Test (FRT) will be used to measure trunk stability during reaching. The amount of lateral stretching will be measured from the tip of the 3rd metacarpal bone in a sitting position and at the edge of the wall.
Trunk Impact Scale | 5 minutes
  Trunk Impact Scale (TIS) will be used to functionally evaluate the trunk in the sitting position. It has three subsections: static and dynamic sitting balance and coordination.
Quality of Upper Extremity Skills Test | 10 minutes
  The Quality of Upper Extremity Skills Test (QUEST) will be used to evaluate the quality of upper extremity skills. The test is a criterion-referenced observational evaluation test consisting of 34 items. It consists of four subsections: "discrete movement", "grip", "weight transfer" and "protective extension". In the heterogeneous movements section of QUEST; The active joint movements of the child's upper extremity are observed one by one and scored according to the items. In the grip section; Functions such as grasping a cube, holding a pencil, grasping a chickpea are evaluated. In the weight transfer section, the child is asked to transfer weight to the front, side and back with his upper extremities while sitting. In the protective extension section, the protective extension reaction of the child forward, sideways and backward in response to a sudden push in a certain direction while the child is sitting is examined.
Constipation Assessment Scale | 2 minutes
  The Constipation Assessment Scale (CAS) will be used to evaluate children's constipation status. This scale evaluates the presence and severity of constipation in children and adults. This scale, consisting of nine questions, is a valid and reliable tool.
Functional Independence Measure for Children | 3 minutes
  Children's functional independence assessments The Functional Independence Measure for Children (WeeFIM) will be used. WeeFIM is a modified version of the Functional Independence Measure (FIM), which was developed for adults, for children. It consists of 6 subheadings, including self-care, sphincter control, transfer, movement, communication and social status, and a total of 18 questions. Scoring is made between 1-7, with a high score defining a good level of functional independence.

SECONDARY OUTCOMES:
Cerebral Palsy Quality of Life Questionnaire | 10 minutes
  The Cerebral Palsy Quality of Life Questionnaire will be used for health-related quality of life assessment. This questionnaire is a scale consisting of child and parent items in 7 areas such as "feelings about function", "participation and physical health".
Selective Control Assessment of the Lower Extremity. | 5 minutes
  Selective Control Assessment of the Lower Extremity (SCALE) will be used to evaluate individuals' lower extremity selective motor control. It is a valid and reliable method in which selective control of lower extremity joint movements is scored between 0-2 points.
Test of Arm Selective Control | 5 minutes
  Test of Arm Selective Control (TASC), developed by Sukal-Moulton et al. in 2017, was used to evaluate children's upper extremity selective motor control. Each movement was scored as 0 (absent), 1 (affected) or 2 (normal) according to descriptive subparameters.
Drooling Impact Scale | 3 minutes
  he Drooling Impact Scale was completed by the same rater on two occasions, 1 month apart, to assess the impact of drooling in children who were expected to be stable. The scale has been shown to behave as expected in validity studies, to have good test-retest reliability in stable children, and to be responsive to change in children who have undergone saliva-control interventions
Pittsburgh Sleep Quality Index | 5 minutes
  It is an index consisting of a total of 24 items that evaluate subsections such as sleep quality and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pennati GV, Bergling H, Carment L, Borg J, Lindberg PG, Palmcrantz S. Effects of 60 Min Electrostimulation With the EXOPULSE Mollii Suit on Objective Signs of Spasticity. Front Neurol. 2021 Oct 15;12:706610. doi: 10.3389/fneur.2021.706610. eCollection 2021. PMID 34721255
- [Result] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Result] Perpetuini D, Russo EF, Cardone D, Palmieri R, De Giacomo A, Pellegrino R, Merla A, Calabro RS, Filoni S. Use and Effectiveness of Electrosuit in Neurological Disorders: A Systematic Review with Clinical Implications. Bioengineering (Basel). 2023 Jun 2;10(6):680. doi: 10.3390/bioengineering10060680. PMID 37370612
- [Result] Bakaniene I, Urbonaviciene G, Janaviciute K, Prasauskiene A. Effects of the Inerventions method on gross motor function in children with spastic cerebral palsy. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):581-586. doi: 10.1016/j.pjnns.2018.07.003. Epub 2018 Jul 20. PMID 30061001